CLINICAL TRIAL: NCT06660407
Title: Grid Radiotherapy for Advanced Non-Small Cell Lung Cancer at the Time of Progression on Immune Checkpoint Inhibition
Brief Title: Grid Radiation Therapy for the Treatment of Stage IV Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMROR2221; NCI-2024-08757 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GMROR2221 (Other: Mayo Clinic); 22-008589 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Specimen Handling; Immunotherapy; Adjuvants, Immunologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (grid radiation therapy) (Experimental): Patients undergo grid radiation therapy over a single fraction on day 1 and palliative radiation therapy over 5 fractions on days 2 and -1 post-grid in the absence of disease progression or unacceptable toxicity. Patients also receive SOC immunotherapy and undergo CT at the discretion of the physician and undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Immunotherapy; Radiation: Palliative Radiation Therapy; Radiation: Spatially-fractionated Radiation Therapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Immunotherapy — Given immunotherapy
  Other Names: Immunological; Immunological Therapy; Immunologically Directed Therapy
Radiation: Palliative Radiation Therapy — Undergo palliative radiation therapy
  Other Names: Palliative Radiotherapy
Radiation: Spatially-fractionated Radiation Therapy — Undergo grid radiation therapy
  Other Names: GRID Therapy; SFRT

SUMMARY:
This phase II trial tests the safety and effectiveness of the combination of grid radiation therapy and standard of care (SOC) immunotherapy in treating patients with stage IV non-small lung cancer (NSCLC). Conventional radiation therapy treatments typically deliver the same radiation dose to the entire tumor. Spatially fractionated radiation therapy or grid therapy is approved and a technique which permits the delivery of high doses of radiation to small regions of the tumor which can lead to enhanced tumor cell killing. Grid therapy has been shown to produce dramatic relief of severe symptoms, significant tumor regression (decrease in the size of a tumor), and above average local control rates often exceeding those expected with conventionally delivered radiation treatments, all with minimal associated toxicity. Immunotherapy has become combined into treating patients, which has led improvements in survival and quality of life. Immunotherapy is now the cornerstone of SOC therapy for stage IV NSCLC. Grid radiation therapy combined with immunotherapy may be safe and effective in treating patients with stage IV NSCLC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To describe the safety and toxicity of grid + immunotherapy in stage IV NSCLC using any Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.

SECONDARY OBJECTIVE:

I. Evaluation of objective response rate using Immune-based Response Evaluation Criteria in Solid Tumors (iRECIST) in non-irradiated lesion(s) after grid therapy in the setting of ongoing immunotherapy.

CORRELATIVE RESEARCH:

I. Monitoring of peripheral blood T cell activation and immunity markers before and after grid therapy.

II. Evaluation of objective response rate using RECIST in the irradiated lesion after grid therapy.

III. Evaluation of time to change in systemic therapy. IV. Evaluation of overall survival.

OUTLINE:

Patients undergo grid radiation therapy over a single fraction on day 1 and palliative radiation therapy over 5 fractions on days 2 and -1 post-grid in the absence of disease progression or unacceptable toxicity. Patients also receive SOC immunotherapy and undergo computed tomography (CT) at the discretion of the physician and undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days then every 8-12 weeks and every 3 months up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) 0, 1, or 2
* Stage IV non-small cell lung cancer progressing on standard of care first line immunotherapy or chemoimmunotherapy
* Patients have not had stereotactic body radiotherapy (SBRT) ≤ 30 days prior to registration
* Extracranial lesion ≥ 3 cm amenable to grid therapy

  * Patients with brain metastases are permitted to enroll if all of the following are true:

    * They are stable (without evidence of progression by imaging ≤ 30 days prior to enrollment and any neurologic symptoms have returned to baseline)
    * Have no evidence of new or enlarging brain metastases, and
    * Are not using steroids ≤ 14 days prior to enrollment
  * Patients may receive conventional palliative radiation to up to 2 other metastatic sites (with at least one evaluable non-irradiated lesion)
* Hemoglobin ≥ 9.0 g/dL (obtained ≤ 15 days prior to enrollment)
* Absolute neutrophil count (ANC) ≥ 1500/mm^3 (obtained ≤ 15 days prior to enrollment)
* Platelet count ≥ 100,000/mm^3 (obtained ≤ 15 days prior to enrollment)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) or direct bilirubin ≤ ULN if total bilirubin is > 1.5 x ULN (obtained ≤ 15 days prior to enrollment)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for patients with liver involvement) (obtained ≤ 15 days prior to enrollment)
* Creatinine ≤ 1.5 x ULN OR glomerular filtration rate (GFR) > 60 mL/min for patients with creatinine > 1.5 x ULN (obtained ≤ 15 days prior to enrollment)
* Negative pregnancy test done ≤ 7 days prior to registration for females of childbearing potential only
* Provide written informed consent
* Willing to provide mandatory blood specimens for correlative research
* Willing to return to Mayo Clinic for follow-up (during the Active Monitoring Phase of the study)
* Estimated by investigator to have a life expectancy > 3 months

Exclusion Criteria:

* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Active autoimmune disease requiring systemic treatment, documented history of severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents

  * NOTE: Exceptions are allowed for:

    * Vitiligo
    * Resolved childhood asthma/atopy
    * Intermittent use of bronchodilators or inhaled steroids
    * Daily steroids at dose of ≤ 10mg of prednisone (or equivalent)
    * Local steroid injections
    * Stable hypothyroidism on replacement therapy
    * Stable diabetes mellitus on non-insulin therapy
    * Sjogren's syndrome
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring systemic therapy
  * Interstitial lung disease
  * Serious, chronic gastrointestinal conditions associated with diarrhea (e.g., Crohn's disease or others)
  * Known active hepatitis B (i.e., known positive hepatitis B virus [HBV] surface antigen [HBsAg] reactive)

    • Known active hepatitis C (i.e., positive for hepatitis C virus [HCV] ribonucleic acid [RNA] detected by polymerase chain reaction [PCR])
  * Known active tuberculosis (TB)
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Unstable cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements (e.g., substance abuse)
* History of myocardial infarction ≤ 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Hypersensitivity to immunotherapy
* Previous adverse event attributed to immunotherapy that led to drug discontinuation
* History of grade 3+ immune-related adverse event or any grade of immune-related neurologic or ocular adverse event while receiving immunotherapy

  * Note: Patients who had endocrine adverse events ≤ grade 2 are allowed to enroll if they are stable on appropriate replacement therapy and asymptomatic
* Other active malignancy < 6 months prior to registration

  * EXCEPTIONS: Non-melanotic skin cancer, papillary thyroid cancer, prostate cancer, or carcinoma-in-situ of the cervix, or others curatively treated and now considered to be at less than 30% risk of relapse
* History of allogenic organ transplantation
* History of active primary immunodeficiency
* Known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice)
* Known active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody (anti-HBc), at screening. Participants with a past or resolved HBV infection (defined as the presence of anti-HBc and absence of HBsAg) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2027-01-10 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
Rate of grade 3+ adverse events | Up to 3 months post-grid treatment
  Will be assessed using any Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Will not utilize a formal statistical design. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be provided. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. Will be considered official if the rate is less than 40% possibly related to study treatment.

SECONDARY OUTCOMES:
Objective response rate | Up to 3 months post-grid treatment
  Will be defined as the number of evaluable patients achieving a response (partial response or better) during treatment with study therapy divided by the total number of evaluable patients. Will be estimated using the Immune-based Response Evaluation Criteria in Solid Tumors in non-irradiated lesion(s) after grid therapy. Point estimates will be generated with 90% confidence intervals using Fisher's exact method. Graphical methods will be used as well, such as waterfall plots.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Owen, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials